CLINICAL TRIAL: NCT03837509
Title: A Randomized Open-Label Phase 1/2 Study of INCB001158 Combined With Subcutaneous (SC) Daratumumab, Compared to Daratumumab SC, in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: INCB001158 Combined With Subcutaneous (SC) Daratumumab, Compared to Daratumumab SC, in Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This decision follows recruitment difficulties. No safety-related concerns impacted this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 01158-206; 2018-004076-35 (EudraCT Number)
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Arginase inhibitor; multiple myeloma; Daratumumab
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: An initial equal randomization of participants between INCB001158 in combination with daratumumab SC (Treatment Group A), daratumumab SC monotherapy (Treatment Group B), and INCB001158 monotherapy (Treatment Group C) will be conducted. Participants in the treatment groups B and C at confirmed disease progression will be crossed over to INCB001158 + daratumumab SC. After the equal randomization period, a response adaptive randomization design will be used to compare the objective response rate of Treatment Groups A and B with adjustments to the randomization rate based on the observed objective response rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- INCB001158 + daratumumab SC (Experimental): INCB001158 + daratumumab
  Interventions: Drug: INCB001158; Biological: Daratumumab SC
- Daratumumab monotherapy and crossover to INC001158+ daratumumab SC (Active Comparator): Daratumumab will be administered as monotherapy, once confirmed disease progression participants will be crossed over to INCB001158+daratumumad combination therapy.
  Interventions: Biological: Daratumumab SC
- INCB001158 monotherapy and crossover to INC001158+ daratumumab SC (Experimental): INCB001158 will be administered as monotherapy, once confirmed disease progression participants will be crossed over to INCB001158+daratumumad combination therapy.
  Interventions: Drug: INCB001158

INTERVENTIONS:
Drug: INCB001158 — Phase 1: INCB001158 administered orally twice daily at the protocol-defined starting dose, with dose escalation/de-escalation based on protocol-defined toxicity criteria to determine the maximum tolerated dose. INCB001158 is administered in combination with daratumumab SC. Phase 2: INCB001158 administered orally at the recommended dose from Phase 1 either as a monotherapy or in combination with daratumumab SC.
  Arms: INCB001158 + daratumumab SC; INCB001158 monotherapy and crossover to INC001158+ daratumumab SC
Biological: Daratumumab SC — Daratumumab 1800 mg co-formulated with rHuPH20 (2000 U/mL) and administered subcutaneously once weekly for Cycles 1 and 2, once every 2 weeks for Cycles 3 to 6, and then once every 4 weeks. Daratumumab will be administered either as monotherapy or in combination with INCB001158.
  Arms: Daratumumab monotherapy and crossover to INC001158+ daratumumab SC; INCB001158 + daratumumab SC

SUMMARY:
The purpose of this study is to evaluate the safety and antitumor activity of INCB001158 in combination with daratumumab SC, compared with daratumumab SC alone, in participants with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of multiple myeloma according to IMWG diagnostic criteria.
* Measurable disease at screening.
* Has received at least 3 but not more than 5 prior lines of multiple myeloma treatment, including proteasome inhibitor, immunomodulatory drug, and anti-CD38 therapies.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Willing to avoid pregnancy or fathering children.
* Willing to provide fresh and archival bone marrow aspiration and biopsy tissue.

Exclusion Criteria:

* Receipt of any of the following treatment within the indicated interval before the first administration of study drug:

  * Anti-myeloma treatment within 2 weeks or 5 half-lives (whichever is longer).
  * Investigational drug (including investigational vaccines) or invasive investigational medical device within 4 weeks.
  * Autologous stem cell transplant within 12 weeks, or allogeneic stem cell transplant at any time.
  * Plasmapheresis within 4 weeks.
  * Radiation therapy within 2 weeks.
  * Major surgery within 2 weeks, or inadequate recovery from an earlier surgery, or surgery planned during the time the participant is expected to participate in the study or within 2 weeks after the last dose of study treatment.
* Toxicity ≥ Grade 2 from previous anti-myeloma therapy except for stable chronic toxicities (≤ Grade 2) not expected to resolve, such as stable Grade 2 peripheral neuropathy.
* Known additional malignancy (other than multiple myeloma) that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry.
* Laboratory values at screening outside the protocol-defined range.
* Significant concurrent, uncontrolled medical condition including but not limited to known chronic obstructive pulmonary disease (COPD), persistent asthma, or history of asthma within the past 2 years; chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment; acute diffuse infiltrative pulmonary disease; clinically significant or uncontrolled cardiac disease.
* Plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome, or amyloidosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Gogov, MD, Study Director — Incyte Corporation
Locations (29):
- United States (14):
  - Southern Cancer Center, Daphne, Alabama
  - Arizona Oncology Associates (Wilmot), Tucson, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada - Twain, Las Vegas, Nevada
  - New York Oncology Hematology, Albany, New York
  - Lineberger Comprehensive Cancer Center At University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Fort Worth South Henderson, Fort Worth, Texas
  - Texas Oncology San Antonio, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists-Fairfax, Fairfax, Virginia
- Germany (4):
  - Charite - Universit�Tsmedizin Berlin, Berlin
  - University of Heidelberg, Heidelberg
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universitatsklinikum Munster, Münster
- Spain (11):
  - Hospital General Universitari Vall D Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Ico Institut Catala D Oncologia, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario Y Politcnico de La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: INCB001158 75 mg BID + Daratumumab: In Phase 1, participants received oral INCB001158 75 milligrams (mg) twice daily (BID) in 28-day cycles starting at Cycle 1, and 1800 mg subcutaneous daratumumab, administered once weekly for Cycles 1 and 2, once every 2 weeks for Cycles 3 to 6, and once every 4 weeks thereafter. Treatment continued until disease progression, unacceptable toxicity, or discontinuation from study treatment for any other reason.
- Phase 1: INCB001158 100 mg BID + Daratumumab; Phase 2: INCB001158 100 mg BID + Daratumumab: In Phase 1, participants received oral INCB001158 100 mg BID in 28-day cycles starting at Cycle 1, and 1800 mg subcutaneous daratumumab, administered once weekly for Cycles 1 and 2, once every 2 weeks for Cycles 3 to 6, and once every 4 weeks thereafter. Treatment continued until disease progression, unacceptable toxicity, or discontinuation from study treatment for any other reason.
- Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab: In Part 1 of Phase 2, participants received daratumumb 1800 mg subcutaneous daratumumab, administered once weekly for Cycles 1 and 2 (28-day cycles), once every 2 weeks for Cycles 3 to 6, and once every 4 weeks thereafter. At the time of confirmed disease progression, participants crossed over to Part 2 of Phase 2 to receive oral INCB001158 100 mg BID starting at Cycle 1, and 1800 mg subcutaneous daratumumab, administered once weekly for Cycles 1 and 2, once every 2 weeks for Cycles 3 to 6, and once every 4 weeks thereafter. Treatment in Phase 2 continued for as long as participants were receiving clinical benefit and did not met any criteria for study withdrawal.
- Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab: In Part 1 of Phase 2, participants received oral INCB001158 100 mg BID in 28-day cycles starting at Cycle 1. At the time of confirmed disease progression, participants crossed over to Part 2 of Part 2 to receive oral INCB001158 100 mg BID starting at Cycle 1, and 1800 mg subcutaneous daratumumab, administered once weekly for Cycles 1 and 2, once every 2 weeks for Cycles 3 to 6, and once every 4 weeks thereafter. Treatment in Phase 2 continued for as long as participants were receiving clinical benefit and did not met any criteria for study withdrawal.
Period: Phase 1
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Started | 6 | 4 | 0 | 0 | 0
Completed | 1 | 2 | 0 | 0 | 0
Not Completed | 5 | 2 | 0 | 0 | 0
Not completed — Death | 5 | 2 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Started | 0 | 0 | 2 | 1 | 2
Disease Progression in Part 1 | 0 | 0 | 0 | 1 | 2
Completed | 0 | 0 | 2 | 0 | 1
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab | Total
Number analyzed (Participants) | 6 | 4 | 2 | 1 | 2 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (11.70) | 68.0 (9.83) | 67.0 (12.73) | NA (NA) — To protect participant privacy, a mean age and standard deviation are not reported for a single participant. | 71.5 (19.09) | 67.1 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | NA — To protect participant privacy, sex is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 4 | 2 | 1 | NA — To protect participant privacy, sex is not reported for a single participant. | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | NA — To protect participant privacy, ethnicity is not reported for a single participant. | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | 6 | 4 | 2 | NA — To protect participant privacy, ethnicity is not reported for a single participant. | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | 0 | NA — To protect participant privacy, ethnicity is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | NA — To protect participant privacy, race is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | 0 | 0 | 0 | NA — To protect participant privacy, race is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | NA — To protect participant privacy, race is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | 1 | 0 | 0 | NA — To protect participant privacy, race is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 5 | 4 | 2 | NA — To protect participant privacy, race is not reported for a single participant. | 2 | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | 0 | 0 | 0 | NA — To protect participant privacy, race is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | 0 | NA — To protect participant privacy, race is not reported for a single participant. | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an adverse event (AE) that was reported for the first time or the worsening of a pre-existing event after the first dose of study treatment.
Time Frame: up to 454 days
Population: Full Analysis Population: all participants enrolled in the study who received at least 1 dose of study treatment (INCB001158 or daratumumab subcutaneous [SC]). Participants were to be analyzed according to the treatment they were assigned to.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab
Number analyzed (Participants) | 6 | 4
Participants | 6 | 4

2. Primary Outcome: Phase 2: Overall Response Rate (ORR): Number of Participants With a Documented Response of Complete Response (CR), Very Good Partial Response (VGPR), or PR, as Per International Myeloma Working Group (IMWG) Criteria
Description: CR: negative immunofixation on serum/urine, disappearance of soft tissue plasmacytomas, <5% bone marrow plasma cells (PCs). VGPR: serum/urine M-component detectable by immunofixation but not on electrophoresis, or ≥90% reduction in serum M-protein (SMP) plus urine M-protein (UMP) <100 milligrams (mg)/24 hours. PR: ≥50% reduction of SMP and reduction in 24-hour UMP by ≥90% or to <200 mg/24 hours. SMP and UMP not measurable: decrease of ≥50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria. SMP and UMP not measurable, and serum free light assay is not measurable: ≥50% reduction in bone marrow PCs is required in place of M-protein, if Baseline bone marrow PC percentage was ≥30%. If present at Baseline, a ≥50% reduction in the size of soft tissue plasmacytomas is required.
Time Frame: up to Day 386
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 2 | 1 | 2
Participants | 0 | 0 | 0

3. Secondary Outcome: Phase 1: ORR: Number of Participants With a Documented Response of CR, VGPR, or PR, as Per IMWG Criteria
Description: as for outcome 2
Time Frame: up to Day 395
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

4. Secondary Outcome: Phase 2: Number of Participants With Any TEAE
Description: A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of study treatment.
Time Frame: up to 420 days
Population: Full Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 2 | 1 | 2
Participants | 1 | 1 | 1

5. Secondary Outcome: Phase 1: Time to Response, Defined as the Time From the First Dose of Study Drug to the First Documented Response of PR or Better (CR, VGPR, or PR), as Per IMWG Criteria
Description: as for outcome 2
Time Frame: up to Day 395
Population: No participants had a response of PR or better; thus, analysis was not conducted.
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 2: Time to Response, Defined as the Time From the First Dose of Study Drug to the First Documented Response of PR or Better (CR, VGPR, or PR), as Per IMWG Criteria
Description: as for outcome 2
Time Frame: up to Day 386
Population: No participants had a response of PR or better; thus, analysis was not conducted.
Arm/Group | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Phase 1: Duration of Response, Defined as Time From First Documented Response of PR or Better (CR, VGPR, PR), as Per IMWG Criteria, Until Date of Disease Progression or Death, Whichever Occurred First
Description: as for outcome 2
Time Frame: up to Day 395
Population: No participants had a response of PR or better; thus, analysis was not conducted.
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase 2: Duration of Response, Defined as Time From First Documented Response of PR or Better (CR, VGPR, PR), as Per IMWG Criteria, Until Date of Disease Progression or Death, Whichever Occurred First
Description: as for outcome 2
Time Frame: up to Day 386
Population: No participants had a response of PR or better; thus, analysis was not conducted.
Arm/Group | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Progression-free Survival (PFS), Defined as the Duration From the Date of the First Dose of Study Drug Until Either Progressive Disease, as Per IMWG Criteria, or Death, Whichever Occurred First
Description: Progressive disease: increase of 25% from the lowest response value in any one of the following: (a) serum M-component (absolute increase must be ≥0.5 grams per deciliter [g/dL]); (b) urine M-component (absolute increase must be ≥200 mg/24 hours); (c) only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/dL); (d) only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell (PC) percentage (absolute percentage must be ≥10%); (d) bone marrow PC percentage: the absolute percentage must be > 10%; (e) definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; (f) development of hypercalcemia (corrected serum calcium > 11.5 mg/dL) that can be attributed solely to the PC proliferative disorder.
Time Frame: up to approximately 2 years
Population: Full Analysis Population. As a result of an early-termination decision following a recruitment challenge (no safety-related concerns), a formal analysis was not performed due to an insufficient number of participants enrolled in Phase 2. PFS was calculated for individual participants, but data were not formally analyzed.
Measure: Number; unit: days
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 6 | 4 | 2 | 1 | 2
days
  Minimum value, uncensored | 8 | 26 | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants.
  Maximum value, uncensored | 337 | 169 | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants.

10. Secondary Outcome: Phase 1: Minimal Residual Disease (MRD), Defined as the Percentage of MRD-negative Participants
Description: Bone marrow aspirate was to be collected for MRD analysis.
Time Frame: up to approximately 2 years
Population: The MRD assay required an analysis to be performed at Baseline and another analysis to be performed at the time of suspected complete response. At the time enrollment was halted, no participants had a complete response; thus, MRD analysis was not performed.
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase 2: MRD, Defined as the Percentage of MRD-negative Participants
Description: Bone marrow aspirate was to be collected for MRD analysis.
Time Frame: up to approximately 2 years
Population: as for outcome 10
Arm/Group | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the first dose of study drug to death from any cause until study completion.
Time Frame: up to 923 days (approximately 2.5 years)
Population: Full Analysis Population. As a result of an early-termination decision following a recruitment challenge (no safety-related concerns), a formal analysis was not performed due to an insufficient number of participants enrolled in Phase 2. Overall survival was calculated for individual participants, but data were not formally analyzed.
Measure: Number; unit: days
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab
Number analyzed (Participants) | 6 | 4 | 1 | 2 | 1
days
  Minimum value, uncensored | 113 | 127 | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants.
  Maximum value, uncensored | 766 | 604 | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants. | NA — Minimum and maximum data values cannot be reported; doing so for the small sample size could lead to the re-identification of participants.

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for up to 454 days; All-cause Mortality was assessed for up to 923 days (approximately 2.5 years).
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events that were reported for the first time or the worsening of pre-existing events after the first dose of study treatment, have been reported.
Groups:
- Total: Total
Arm/Group | Phase 1: INCB001158 75 mg BID + Daratumumab | Phase 1: INCB001158 100 mg BID + Daratumumab | Phase 2: INCB001158 100 mg BID + Daratumumab | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab | Total
All-Cause Mortality (participants affected / at risk) | 5/6 | 2/4 | 0/2 | 1/1 | 1/2 | 9/15
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/4 | 0/2 | 1/1 | 0/2 | 5/15
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 1/2 | 1/1 | 1/2 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: INCB001158 75 mg BID + Daratumumab (N=6) | Phase 1: INCB001158 100 mg BID + Daratumumab (N=4) | Phase 2: INCB001158 100 mg BID + Daratumumab (N=2) | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab (N=1) | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab (N=2) | Total (N=15)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: INCB001158 75 mg BID + Daratumumab (N=6) | Phase 1: INCB001158 100 mg BID + Daratumumab (N=4) | Phase 2: INCB001158 100 mg BID + Daratumumab (N=2) | Phase 2: Daratumumab Monotherapy; Cross Over to INCB001158 + Daratumumab (N=1) | Phase 2: INCB001158 Monotherapy; Cross Over to INCB001158 + Daratumumab (N=2) | Total (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dysstasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Listless (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oroticaciduria (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
The study was terminated following a recruitment challenge. There were no safety-related concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03837509/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03837509/SAP_001.pdf